CLINICAL TRIAL: NCT02752360
Title: Biodegradable Stenting Anastomoses Versus Double-layer Hand Sutures for Reconstruction in Surgery of Intestinal Anastomosis: A Multicenter, Prospective Cohort Study
Brief Title: Biodegradable Stenting Anastomoses Versus Double-layer Hand Sutures for Reconstruction in Intestinal Anastomosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Doctor, Beijing Friendship Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BjFH20160410-1
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Colonic Neoplasms; Diverticulosis, Colonic; Crohn Disease
Keywords: intestinal reconstruction; end to end anastomosis
MeSH Terms: conditions — Colonic Neoplasms; Diverticulosis, Colonic; Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BSA Group (Experimental): Patients accept the management of Biodegradable Stenting Anastomoses for reconstruction in the surgery of Intestinal Anastomosis
  Interventions: Procedure: Biodegradable Stenting Anastomoses
- DHS Group (Experimental): Patients accept the management of Double-layer Hand Sutures for reconstruction in the surgery of Intestinal Anastomosis
  Interventions: Procedure: Double-layer Hand Sutures

INTERVENTIONS:
Procedure: Biodegradable Stenting Anastomoses — Biodegradable Stenting Anastomoses(BSA) is a new method and device which helps to make intestinal anastomosis easily. According to the measurement of intestinal canal diameter, chose an appropriate size of BSA and use the Seromuscular layer Purse-string Suture to stitch with an absorbable line (VCP311, Ethicon, Inc.) away from the end 0.5 to 1.0 cm and not knot temporarily, then open and sterilize intestinal canal fully, and place the BSA into the intestinal canal at appropriate position before tightening knot. Last, the interrupted whole layer inversion suture is used to fix.
  Arms: BSA Group
Procedure: Double-layer Hand Sutures — Double-layer Hand Sutures(DHS)is a surgery way that is to use the single-layer continous Hand Sutures,then Lembert to stitch with an absorbable line (VCP311, Ethicon, Inc.).
  Arms: DHS Group

SUMMARY:
Intestinal anastomosis plays an important role in various general surgeries, but the complications such as anastomotic leakage,stenosis and hemorrhage cannot been avoided. Although many ways are put up to solve this problem, there are still many imports need to improve. Therefore, the Biodegradable Stenting Anastomoses(BSA), which make intestinal anastomosis easily and less complications, have been produced.The major goal of this study is to evaluate the efficacy of Biodegradable Stenting Anastomoses(BSA) for reconstruction in surgery of intestinal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 - 80 years.
* Patients with operation of end to end anastomosis of colon or small intestine.
* Patients without previous surgery during 3 months.
* Patients who understand the nature of this trial and provide informed consent.

Exclusion Criteria:

* Patients with severe cardiopulmonary disease or other severe disease.
* Patients who are psychopath, pregnant, and child without capacity for civil conduct.
* Patients with complete intestinal obstruction.
* Patients with abdominal cavity infection.
* Patients who are treating by drug such as adrenal cortical hormone and immune inhibitors, chemotherapy drugs, radiation and so on.
* Patients who need to accept the anastomosis between rectum and colon.
* Patients who are required to accept intestinal anastomosis twice or more.
* Patients who are required to accept the treatment of colostomy.
* other conditions that render a patient unsuitable for the trial as determined by the study investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leakage Rate | 7-10 Days
  The patients with anastomotic leakage / the total patients. The definition of anastomotic leakage in this study, is included one of the situation as follows: (1) peritonitis caused by leakage, pelvic abscess without radiologically proven anastomotic leakage were considered as equivalents of clinically anastomotic leakage as defined above.; (2) Discharge of faeces, pus or gas from the abdominal drain; (3) All anastomotic leakages were confirmed by one or more of the following methods such as CT scan, ultrasonography and laparotomy.
Anastomotic Hemorrhage Rate | 2 Weeks
  The patients with anastomotic hemorrhage / the total patients. Anastomotic bleeding was considered gastrointestinal bleeding after surgery, and it ascertains that the bleeding is from anastomosis with endoscopy.
Anastomotic Stenosis Rate | 6 Months
  The patients with anastomotic stenosis / the total patients.Anastomotic stenosis which is not caused by tumor in the patients with complete or incomplete intestinal obstruction symptoms.

SECONDARY OUTCOMES:
Number of participant with abnormal laboratory values | 6 Months
  Number of participant with abnormal laboratory values will be record. Laboratory tests include Blood routine/Coagulation/Liver and renal function/Electrolyte/Lipids/OB. Abnormal laboratory values means that values of Laboratory tests beyond the normal values.
Severe adverse events (SAEs) | 6 Months
  Severe adverse events (SAEs) refer to the following conditions: death, life-threatening or permanent or significant disability, permanent functional injury to the organs, hospitalization for emergencies or prolonged hospitalization
Whether the Biodegradable Stenting Anastomoses be eliminated or not | 6 Months
  The enteroscopy will be used to observe whether the Biodegradable Stenting Anastomoses be eliminated from body at 4th weeks after surgery.If Biodegradable Stenting Anastomoses be eliminated, contrast will be filling defect.
The time of reconstruction in the surgery of Intestinal Anastomosis | 1 Day
  The time of reconstruction in the surgery of Intestinal Anastomosis for each group is recorded, which is from the beginning to the ending of Intestinal Anastomosis

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Doctor, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China